CLINICAL TRIAL: NCT02879162
Title: A Phase II Study of Durvalumab and Tremelimumab in Patients With Advanced Rare Tumours
Brief Title: Durvalumab and Tremelimumab in Patients With Advanced Rare Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I228
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced Rare Tumours
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab (Experimental): Durvalumab 1500 mg IV 60 min Day 1 every 4 weeks Tremelimumab 75 mg IV 60 min Day 1, cycles 1-4
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab
Drug: Tremelimumab

SUMMARY:
The standard or usual treatment for this disease may be chemotherapy or other types of treatment to slow the spread of the disease and relieve some symptoms of this cancer.

DETAILED DESCRIPTION:
Durvalumab is a new type of drug for many types of cancer. Laboratory tests show that it works by allowing the immune system to detect cancer and stimulate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals and has been studied in 5000 people and seems promising but it is not clear if it can offer better results than standard treatment alone.

Tremelimumab is a new type of drug for various types of cancers. It works in a similar way to durvalumab and may improve the effect of durvalumab. This may also help slow the growth of the cancer cells or may cause cancer cells to die. Tremelimumab has been shown to shrink tumours in animals and has been studied in 1500 people and seems promising but it is not clear if it can offer better results than standard treatment alone when used with durvalumab

Combinations of durvalumab and tremelimumab have also been studied and when combined have been shown to increase tumour shrinkage in animals compared to either drug alone. While the combination has been studied in 250 people, it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed cancer that is advanced / metastatic / recurrent or unresectable and for which no curative therapy exists as follows:

  1. Salivary carcinoma (excluding adenoid cystic carcinoma histology)
  2. Carcinoma of unknown primary with tumour infiltrating lymphocytes (TILs) and/or expressing PD-L1
  3. Mucosal melanoma
  4. Acral melanoma
  5. Osteosarcoma
  6. Undifferentiated pleomorphic sarcoma
  7. Clear cell carcinoma of the ovary
  8. Squamous cell carcinoma of the anal canal (SCCA)
* All patients must have a tumour tissue from their primary or metastatic tumour available
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to registration (within 35 days if negative).

All patients must have at least one measurable lesion as defined by RECIST 1.1 that has not been the site of the protocol mandated biopsy. The criteria for defining measurable disease are as follows:

CT scan (with slice thickness of 5 mm) ≥ 10 mm --> longest diameter Lymph nodes by CT scan ≥ 15 mm --> measured in short axis

* Patients must be ≥ 16 years of age.
* Patients must have an ECOG performance status of 0 or 1.
* Previous Therapy

Cytotoxic Chemotherapy:

Patients may have received prior chemotherapy - no limit on number of prior regimens.

Other Systemic Therapy:

Patients may have received other prior therapies including, angiogenesis inhibitors, PARP inhibitors or signal transduction inhibitors (tyrosine kinase inhibitors). Prior therapy with PD-1/PD-L1 or CTLA-4 inhibitors is not allowed.

Patients must have recovered from all reversible toxicity related to prior chemotherapy or systemic therapy (unless grade 1, irreversible, or considered by investigator as not clinically significant) and have adequate washout as follows:

Longest of one of the following:

* Two weeks
* 5 half-lives for investigational agents
* Standard cycle length of standard therapies

Radiation:

Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of registration. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG senior investigator. Concurrent radiotherapy is not permitted. Patients planned for concurrent chemotherapy-radiation are not eligible.

Surgery:

Previous surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of registration, and that wound healing has occurred.

* Lab Requirements:

Absolute neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 90 g/L Bilirubin ≤ 1.5 x ULN (upper limit of normal)* AST and ALT ≤ 2.5 x ULN (if liver metastases are present, ≤ 5 x ULN) Serum creatinine < 1.25 x ULN or: Creatinine clearance ≥ 40 mLs/min

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre.
* Subjects should not donate blood while participating in this study, or for at least 90 days following the last infusion of durvalumab or tremelimumab.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient registration

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other cancers curatively treated with no evidence of disease for ≥ 5 years.
* Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia.
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years).
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of registration.
* Live attenuated vaccination administered within 30 days prior to registration.
* History of hypersensitivity to durvalumab or tremelimumab or any excipient. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF ≥ 50%.
* Untreated symptomatic brain metastases or brain metastases in whom radiation or surgery is indicated.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol (incl corticosteroid administration), or would put the patient at risk. This includes but is not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or tuberculosis or any infection requiring systemic therapy).
  * Active peptic ulcer disease or gastritis.
  * Known pneumonitis or pulmonary fibrosis with clinically significant impairment of pulmonary function.
* Pregnant or lactating women.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abha Gupta, Study Chair — Hospital for Sick Children, Toronto ON Canada
Locations (13):
- Canada (13):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta AA, Tinker A, Jonker D, Jamal R, Hirte H, Winquist EW, Chu Q, Kollmannsberger C, Wong R, Alcindor T, Nielsen TO, Tsao M, Cottrell TR, Provencher D, Hilton J, Krzyzanowska MK, Elser C, Hotte S, Sederias J, Zhang S, Tu W, Dancey J. Durvalumab and tremelimumab in patients with advanced rare cancer: a multi-centre, non-blinded, open-label phase II basket trial. EClinicalMedicine. 2024 Dec 10;79:102991. doi: 10.1016/j.eclinm.2024.102991. eCollection 2025 Jan. PMID 39737219

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab + Tremelimumab: Durvalumab 1500 mg IV 60 min Day 1 every 4 weeks Tremelimumab 75 mg IV 60 min Day 1, cycles 1-4
  Durvalumab
  Tremelimumab
Period: Overall Study
Arm/Group | Durvalumab + Tremelimumab
Started | 140
Completed | 138 (Not completed is defined as not treated here.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 138
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.4 [50.6 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 135
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Measured by RECIST Version 1.1
Description: Objective response rate is defined as the proportion of response evaluable patients who had complete response (CR) or partial response (PR) as their best response as assessed by RECIST version 1.1 criteria (i.e. a 30% decrease in the sum of the longest diameters of the target lesions maintained for at least 4 weeks (CR), or complete disappearance of disease and cancer related symptoms, also maintained for at least 4 weeks (CR)).
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 136
Participants
  CR | 1
  PR | 19
  SD | 32
  PD | 76
  IN | 8

2. Secondary Outcome: Time to Progression Based on Kaplan-Meier Method
Description: defined as time from the date of randomization to the date of progression
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 136
months | 2.8 [2.6 to 2.9]

3. Secondary Outcome: Progression Free Survival Based on Kaplan-Meier Method
Description: defined as time from the date of randomization to the date of progression or death
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 136
months | 2.8 [2.6 to 2.8]

ADVERSE EVENTS:
Time Frame: Continuously measured at baseline, day 1 of each cycle, and as clinically indicated, 4 week after completion of protocol therapy, every three months thereafter to follow adverse events felt related until resolved to ≤ Grade 2, to 48 months.
Arm/Group | Durvalumab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 114/138
Serious Adverse Events (participants affected / at risk) | 80/138
Other Adverse Events (participants affected / at risk) | 137/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab + Tremelimumab (N=138)
Diarrhea (Gastrointestinal disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Colitis (Gastrointestinal disorders) | 8
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 6
Immune system disorders - Other specify (Immune system disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 4
Fever (General disorders) | 4
Small intestinal obstruction (Gastrointestinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 2
Fatigue (General disorders) | 2
Infections and infestations - Other specify (Infections and infestations) | 2
Pain (General disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Skin infection (Infections and infestations) | 2
Thromboembolic event (Vascular disorders) | 2
Abdominal infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - Other specify (Cardiac disorders) | 1
Cecal hemorrhage (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Device related infection (Infections and infestations) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Edema limbs (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 1
Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipase increased (Investigations) | 1
Lung infection (Infections and infestations) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Nervous system disorders - Other specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Sudden death NOS (General disorders) | 1
Syncope (Nervous system disorders) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
White blood cell decreased (Investigations) | 1
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab + Tremelimumab (N=138)
Fatigue (General disorders) | 109
Diarrhea (Gastrointestinal disorders) | 64
Nausea (Gastrointestinal disorders) | 61
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 61
Anorexia (Metabolism and nutrition disorders) | 59
Constipation (Gastrointestinal disorders) | 57
Cough (Respiratory, thoracic and mediastinal disorders) | 53
Abdominal pain (Gastrointestinal disorders) | 47
Pruritus (Skin and subcutaneous tissue disorders) | 43
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 42
Back pain (Musculoskeletal and connective tissue disorders) | 40
Vomiting (Gastrointestinal disorders) | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31
Headache (Nervous system disorders) | 29
Hypothyroidism (Endocrine disorders) | 28
Edema limbs (General disorders) | 28
Pain (General disorders) | 28
Insomnia (Psychiatric disorders) | 27
Peripheral sensory neuropathy (Nervous system disorders) | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Fever (General disorders) | 22
Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 21
Dry mouth (Gastrointestinal disorders) | 19
Dizziness (Nervous system disorders) | 19
Hot flashes (Vascular disorders) | 18
Flu like symptoms (General disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 14
Non-cardiac chest pain (General disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Thromboembolic event (Vascular disorders) | 13
Upper respiratory infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 12
Anxiety (Psychiatric disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 12
Sinus tachycardia (Cardiac disorders) | 11
Dysphagia (Gastrointestinal disorders) | 11
Dysgeusia (Nervous system disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 11
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 10
Hyperthyroidism (Endocrine disorders) | 9
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 9
Mucositis oral (Gastrointestinal disorders) | 9
Nervous system disorders - Other specify (Nervous system disorders) | 9
Dry eye (Eye disorders) | 8
Eye disorders - Other specify (Eye disorders) | 8
Bloating (Gastrointestinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 7
Chills (General disorders) | 7
General disorders and administration site conditions - Other specify (General disorders) | 7
Urinary frequency (Renal and urinary disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7
Rectal pain (Gastrointestinal disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal and connective tissue disorder - Other specify (Musculoskeletal and connective tissue disorders) | 6
Paresthesia (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 6
Depression (Psychiatric disorders) | 6
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 6
Lymphedema (Vascular disorders) | 6
Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 5
Blurred vision (Eye disorders) | 5
Rectal hemorrhage (Gastrointestinal disorders) | 5
Immune system disorders - Other specify (Immune system disorders) | 5
Infections and infestations - Other specify (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Confusion (Psychiatric disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Edema face (General disorders) | 4
Allergic reaction (Immune system disorders) | 4
Bruising (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Neuralgia (Nervous system disorders) | 4
Pelvic pain (Reproductive system and breast disorders) | 4
Vaginal discharge (Reproductive system and breast disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 3
Adrenal insufficiency (Endocrine disorders) | 3
Cushingoid (Endocrine disorders) | 3
Conjunctivitis (Eye disorders) | 3
Eye pain (Eye disorders) | 3
Floaters (Eye disorders) | 3
Colitis (Gastrointestinal disorders) | 3
Lung infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Dysphasia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 3
Reproductive system and breast disorders - Other specify (Reproductive system and breast disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 3
Ear pain (Ear and labyrinth disorders) | 2
Watering eyes (Eye disorders) | 2
Anal pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 2
Edema trunk (General disorders) | 2
Infusion related reaction (General disorders) | 2
Localized edema (General disorders) | 2
Rhinitis infective (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Injury poisoning and procedural complications - Other specify (Injury, poisoning and procedural complications) | 2
Wound complication (Injury, poisoning and procedural complications) | 2
Aspartate aminotransferase increased (Investigations) | 2
Cholesterol high (Investigations) | 2
Investigations - Other specify (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 2
Phantom pain (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Vaginal pain (Reproductive system and breast disorders) | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hematoma (Vascular disorders) | 2
Vascular disorders - Other specify (Vascular disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Endocrine disorders - Other specify (Endocrine disorders) | 1
Eyelid function disorder (Eye disorders) | 1
Flashing lights (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Facial pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Injection site reaction (General disorders) | 1
Irritability (General disorders) | 1
Malaise (General disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Infective myositis (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 1
CPK increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
Weight loss (Investigations) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Movements involuntary (Nervous system disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02879162/Prot_SAP_000.pdf